CLINICAL TRIAL: NCT05906706
Title: An Open-Label, Expanded Access Program of Dupilumab in Adult Patients With Bullous Pemphigoid
Brief Title: Compassionate Use of Dupilumab for Adult Patients With Bullous Pemphigoid
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-BP-2290-EAP
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Bullous Pemphigoid
Keywords: Skin Diseases; Autoimmune Diseases; Immune System Diseases; Inflammatory Diseases
MeSH Terms: conditions — Pemphigoid, Bullous; Skin Diseases; Autoimmune Diseases; Immune System Diseases | interventions — dupilumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: dupilumab — Subcutaneous (SC) administration
  Other Names: REGN668; DUPIXENT®; SAR231893

SUMMARY:
The objective of the program is to provide patients with Bullous Pemphigoid (BP), that participated in the R668-BP-1902 (NCT04206553) phase 2/3 study, dupilumab treatment and evaluate the long-term safety of dupilumab.

DETAILED DESCRIPTION:
Expanded Access requests are only being considered in response to intermediate size patient population applications. Availability will depend on location.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completion of the end of study (EOS) visit in the parent dupilumab phase 2/3 study, R668-BP-1902 (NCT04206553)

Key Exclusion Criteria:

1. Patients who, during the parent dupilumab study, R668-BP-1902 (NCT04206553), developed a serious adverse event (SAE) and/or adverse event (AE) deemed related to program drug and which led to discontinuation of investigational product
2. Treatment with non-steroidal immunosuppressive/immunomodulating drug(s) (eg, mycophenolate mofetil, azathioprine, or methotrexate) within 4 weeks before the baseline visit
3. Treatment with BP-directed biologics, as defined in the protocol
4. Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit
5. Planned or anticipated use of any prohibited medications or procedures during program treatment
6. Severe concomitant illness(es) that, in the treating physician's judgment, would adversely affect the patient's participation in the program

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult